CLINICAL TRIAL: NCT06438159
Title: Impact of Mindfulness-Based Stress Reduction Meditation Practice on Medium- and Long-term Follow-up of Cardiac Patients After Cardiac Rehabilitation.
Brief Title: Impact of Mindfulness-Based Stress Reduction Meditation Practice on Patients After Cardiac Rehabilitation.
Acronym: CARDIO-MBSR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CARDIO-MBSR
Record Dates: First submitted 2024-05-23; First posted 2024-05-31 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Cardiac Disease
Keywords: cardiac rehabilitation; MBSR
MeSH Terms: conditions — Heart Diseases | interventions — Cardiac Rehabilitation; Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cardiac rehabilitation with Mindfulness-Based Stress Reduction (MBSR) (Experimental): Conventional cardiac rehabilitation over 4 weeks with the introduction of MBSR over 8 weeks
  Interventions: Other: Cardiac rehabilitation with Mindfulness-Based Stress Reduction (MBSR)
- Conventional cardiac rehabilitation (Active Comparator): Conventional cardiac rehabilitation over 4 weeks
  Interventions: Other: Conventional cardiac rehabilitation

INTERVENTIONS:
Other: Cardiac rehabilitation with Mindfulness-Based Stress Reduction (MBSR) — The MBSR program is as follows:
  * 8 weekly group sessions of 2h30 led by the mindfulness instructor,
  * Sessions of around 45 minutes a day to be carried out by the patient, at home, for personal training,
  * An intensive day between the 6th and 7th sessions to explore certain practices more intensively, in order to support participants in effectively integrating mindfulness meditation into various life situations.
  Arms: Cardiac rehabilitation with Mindfulness-Based Stress Reduction (MBSR)
Other: Conventional cardiac rehabilitation — The usual cardiac rehabilitation program combines exercise training and therapeutic education workshops, with a daily session for four weeks.
  Arms: Conventional cardiac rehabilitation

SUMMARY:
Cardiac rehabilitation is a major component of treatment for patients suffering from coronary pathology revealed by myocardial infarction or acute coronary syndrome warranting transluminal coronary angioplasty, as well as in the aftermath of cardiac surgery.

A significant proportion of patients in this situation (40%) suffer from varying degrees of anxiety and depression, which are difficult to treat. These impair their quality of life and can make it more difficult for them to take part in the rehabilitation program, compromising the results that can be expected. Finally, they are often associated with lax compliance with medical treatment, less control of risk factors and less regular exercise.

Cardiac rehabilitation teams are well aware of this anxiety-depressive picture, and various therapies such as sophrology, relaxation and yoga have been proposed as alternatives to conventional medical treatments to help patients through this period.

Among these alternatives is the concept of "Mindfulness-Based Meditation", based on the Mindfulness-Based Stress Reduction (MBSR) protocol described by Dr. JKabat Zinn.

It has been the subject of several prospective randomized studies, which have demonstrated that it is suitable for the management of patients in this situation, and that it has measurable beneficial effects on their sense of well-being.

To our knowledge, the MBSR program used in cardiac rehabilitation has never been the subject of a randomized comparative study in France to assess its effectiveness on medium- and long-term anxiety-depressive disorders. This is the objective of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Cardiac patients eligible for cardiac rehabilitation,
2. Patient with a Hospital Anxiety and Depression Scale (HADS) score for the anxiety dimension (HADS-A) >7 or a score for the depression dimension (HADS-D) > 7
3. Age ≥ 18 years
4. Affiliated with a social security scheme or beneficiary of such a scheme
5. Patient signed free and informed consent form

Exclusion Criteria:

1. Patients already treated for severe psychiatric disorders (major depression, psychosis, schizophrenia)
2. Inability to follow the 8-week MBSR program
3. Protected patient: minor, adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
4. Medical conditions which may interfere with the conduct of the study and the investigator's judgment, and which may render the patient unfit to participate in the study.
5. Pregnant or breast-feeding patient
6. Refusal to participate in the study or inability to comply with the study protocol for any reason whatsoever

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-11-12 (Estimated); Study Completion 2026-11-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of HADS anxiety and depression scores | Baseline and 12 months
  HADS (Hospital Anxiety and Depression Scale) is a self questionnaire including 14 items which identifies and quantifies the depression and anxiety from which a person suffers.

SECONDARY OUTCOMES:
To assess the quality of life | Baseline, 1 month, 6 months and 12 months
  The patients' quality of life will be measured by the MQOL-R questionnaire, which is a 14-point tool forming 4 subscales: physical, psychological, existential and social.
Medical treatment compliance | Baseline, 1 month, 6 months and 12 months
  The patients' compliance to their medical treatment will be measured by the GIRERD self-questionnaire including 6 questions, to assess compliance, i.e. whether treatment is taken regularly and as prescribed.
Changes from baseline of cardiac risk factor "fasting blood glucose" | Baseline, 1 month, 6 months and 12 months
  fasting blood glucose (in g/L)
Changes from baseline of cardiac risk factor "glycosylated hemoglobin" | Baseline, 1 month, 6 months and 12 months
  glycosylated hemoglobin (% of total hemoglobin)
Changes from baseline of cardiac risk factor "Lipid profile LDLc" | Baseline, 1 month, 6 months and 12 months
  Low Density Lipoprotein cholesterol (g/l)
  * Tobacco consumption (in packs.year)
  * BMI
  * Ricci Gagnon scale and 6-minute walk test
Changes from baseline of cardiac risk factor "Lipid profile HDLc" | Baseline, 1 month, 6 months and 12 months
  High Density Lipoprotein cholesterol (g/l)
Changes from baseline of cardiac risk factor "BMI" | Baseline, 1 month, 6 months and 12 months
  BMI ( weight and height will be combined to report BMI in kg/m2)
Changes from baseline of cardiac risk factor "effort" | Baseline, 1 month, 6 months and 12 months
  6-minute walk test
Changes from baseline of cardiac risk factor "activity" | Baseline, 1 month, 6 months and 12 months
  Ricci Gagnon scale: self questionnaire including 9 questions to evaluate if the subject has an inactive, active or very active profile
Changes from baseline of cardiac risk factor "Tobacco consumption" | Baseline, 1 month, 6 months and 12 months
  Tobacco consumption (in packs.year)
Changes from baseline of cardiac risk factor "Blood pressure measurement" | Baseline, 1 month, 6 months and 12 months
  Blood pressure
To assess the patient's anxiety | Baseline, 1 months and 6 months
  HADS anxiety score
To assess the patient's depression | Baseline, 1 months and 6 months
  HADS depression score
To evaluate the continuation of formal and informal mindfulness meditation practices in patients who have benefited from the MBSR program. | 3 months, 6 months and 12 months
  Patients of the MBSR group will be asked two questions :
  "Do you still do formal meditation practices?" "Do you still do informal meditation practices?"
To evaluate the patient's "mindfulness" and its impact on vital aspects in patients who have benefited from the MBSR program. | 3 months, 6 months and 12 months
  FFMQ (Five Facets Mindfulness Questionnaire) questionnaire, which includes 39 questions, which assess the 5 facets which constitute mindfulness as a construct:
  * Describe the experience: talk about the experience in words.
  * Acting mindfully: performing actions with active attention to each step.
  * Non-judgment: absence of positive or negative comments on the thoughts and emotions experienced.
  * Non-reactivity to private events: allowing thoughts and emotions to exist without responding to them automatically.
  * Observation: remaining aware and focused on the experience, even when it is aversive or painful.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique d'Aressy, Aressy, France

IPD SHARING:
Plan to Share IPD: No